CLINICAL TRIAL: NCT05616546
Title: Longitudinal Analysis of Bone Marrow and Peripheral Blood Immune Responses to Influenza Vaccination in a Healthy Adult Cohort
Brief Title: Bone Marrow and Peripheral Blood Immune Responses Study
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Edmund Waller, Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY00003852; 75N93021C00017 (Other Grant/Funding Number: NIH NATL INST OF ALLERGY AND INFECTIOUS)
Record Dates: First submitted 2022-10-21; First posted 2022-11-15 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Influenza
Keywords: Influenza Vaccine; Bone Marrow; Immune Response
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Influenza Vaccine (Experimental): Healthy male and female individuals aged 18-64 years will be eligible to participate in this study.
  Subjects will be offered the opportunity to participate in the study for up to 3 consecutive years, provided eligibility criteria are met each year. Subjects will be re-screened to verify continued eligibility and re-consented prior to subsequent participation and will receive new subject identifiers
  Interventions: Biological: Influenza Vaccine

INTERVENTIONS:
Biological: Influenza Vaccine — The vaccine used in this study will be a licensed seasonal inactivated influenza vaccine for intramuscular injection that is approved by the FDA. Enrolled subjects will receive licensed seasonal inactivated influenza vaccine (administered as a part of the study).

SUMMARY:
The purpose of this study is to evaluate the immune response of the killed flu vaccine in healthy subjects. Participants in this study are considered to be healthy volunteers. Influenza ("Flu") infection carries a risk of serious illness.

This is an open label and single arm observational study designed to assess the humoral response to influenza vaccination and the longevity of humoral immunity to influenza vaccination in healthy adults.

Enrolled subjects will receive licensed seasonal inactivated influenza vaccine (administered as a part of the study). Participants will donate serial samples of blood and bone marrow aspirate for immunology monitoring. Repeated measurements of humoral immunity will be obtained at 7 days, 28 days, 90 days and at one year post vaccination to assess the magnitude, clonal diversity and persistence of B-cell responses to influenza vaccination.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the immune response of the killed flu vaccine in healthy subjects. Participants in this study are considered to be healthy volunteers. Influenza ("Flu") infection carries a risk of serious illness. The immune system is the body's defense against all kinds of infections and foreign invaders. The flu vaccine is a dose of killed (inactivated) flu virus. The immune system then builds protective responses against the flu virus. These responses help attack and kill the virus. One may not get sick at all, or may have a much shorter or milder illness.

The killed flu vaccine is made from a killed influenza virus that has been split apart and modified in such a way as to not be able to grow at all in humans. The killed flu vaccine is given via an injection into your arm. The purpose of this research study is to test the immune response to a vaccination for influenza (the "flu"). Participants will be given one dose of an FDA-approved influenza vaccine. The flu vaccine used in this study is the same seasonal flu vaccine that is approved by the government for this year.

The study will measure immune response to the seasonal flu vaccine by measuring the immune response in the blood and bone marrow over a period of time, for up to 1 year post (after) vaccination. Researchers expect to see a change in the immune system in response to the flu vaccination. This response will be evaluated by comparing data obtained before flu vaccination to data collected at specified time points (0, 7, 28, 90, and 365 days) after the administration of the flu vaccine. It is possible that by measuring these differences, especially in the bone marrow, clinicians can better understand how the body responds to flu vaccination and how long the immunity lasts. This is important because it could help lead to the creation of more effective flu vaccines in the future.

Up to 90 healthy volunteers will be enrolled into the study. Subjects chosen to participate in this study will be healthy volunteers who are eligible to receive the flu vaccine. An individual's study participation will last for up to 365 days, or 1 year. Subjects who complete the study will be given the option to re-enroll if they meet enrollment criteria. The duration for this study is seven years.

This single site study will take place at Emory University. As this is a healthy volunteers study, flyers, social media posts, and electronic newsletter advertisements will be used to recruit participants for this study. Interested individuals can contact the study team to determine eligibility. We will not request any waivers of consent.

Participants will be asked, as part of the informed consent process, whether or not they agree to have their specimens used only for future research. This decision can be changed at any time by the participant without penalty. Participants who agree to take part in this study will have specimens collected for antibody determination and viral typing. Each specimen will be labeled only with a unique tracking number to protect participant's confidentiality. These samples will not be used for genetic (DNA) studies and will be stored in a coded manner indefinitely.

ELIGIBILITY:
Inclusion Criteria:

* All genders, races and ethnic groups (inclusive of women and minorities) are eligible for this trial, as influenza and the associated range of clinical issues accompanying influenza infection can impact people of all genders, races and ethnic groups. It is anticipated that the distribution of study participants will be diverse with regard to these demographics.
* Adults able to provide consent on their own
* Healthy adults

Exclusion Criteria:

* Adults unable to consent
* Women who are pregnant or nursing a child may not take part in this study. If a woman of childbearing potential is enrolled in this study, she and the study doctor must agree on a method of birth control to use throughout the study. Enrollees who think that they may have gotten pregnant during the study must tell the study doctor immediately. Pregnant women will be taken out of the study.
* Prisoners
* Cognitively impaired or individuals with impaired decision-making capacity
* Individuals who are vulnerable to coercion or undue influence (human fetuses, or neonates of uncertain viability or non-viable neonates, minors/children, and cognitively impaired adults) will not be eligible for participation in this study.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-10-16 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Changes in clonal diversity of B-Cell response to Influenza in blood | Study Days: 0, 7, 28, 90, 365
  Blood samples will be drawn, labeled, and logged at the Georgia Clinical & Translational Science Alliance (CTSA) of Emory University by a skilled clinical research nurse or phlebotomist. Blood samples will be drawn and stored in 8ml CPT tubes. These samples will be maintained at room temperature until they are transported to the laboratory.
  Clonal diversity of B-Cell response to Influenza in blood will be measured on study days 0, 7, 28, 90, and 365, and compared for changes.
Changes in clonal diversity of B-Cell response to Influenza in bone marrow | Study Days 0, 28, 365
  Bone marrow aspirate specimens will be drawn, labeled, and logged at the Georgia Clinical & Translational Science Alliance (CTSA) by the Principal Investigator. These samples will be collected in 10 ml sodium heparin tubes and labeled with coded subject information. They will be maintained at room temperature until they are transported to the laboratory.
  Clonal diversity of B-Cell response to Influenza in bone marrow, will be measured on study days 0, 28, and 365, and compared for changes.
Changes in magnitude of B-Cell response to Influenza in blood | Study Days: 0, 7, 28, 90, 365
  Blood samples will be drawn, labeled, and logged at the Georgia Clinical & Translational Science Alliance (CTSA) of Emory University by a skilled clinical research nurse or phlebotomist. Blood samples will be drawn and stored in 8ml CPT tubes. These samples will be maintained at room temperature until they are transported to the laboratory.
  Magnitude of B-Cell response to Influenza will be measured on study days 0, 7, 28, 90, and 365, and compared for changes.
Changes in magnitude of B-Cell response to Influenza in bone marrow | Study Days 0, 28, 365
  Bone marrow aspirate specimens will be drawn, labeled, and logged at the Georgia Clinical & Translational Science Alliance (CTSA) by the Principal Investigator. These samples will be collected in 10 ml sodium heparin tubes and labeled with coded subject information. They will be maintained at room temperature until they are transported to the laboratory.
  Magnitude of B-Cell response to Influenza in bone marrow, will be measured on study days 0, 28, and 365, and compared for changes.
Changes in persistence of B-Cell response to Influenza in blood | Study Days: 0, 7, 28, 90, 365
  Blood samples will be drawn, labeled, and logged at the Georgia Clinical & Translational Science Alliance (CTSA) of Emory University by a skilled clinical research nurse or phlebotomist. Blood samples will be drawn and stored in 8ml CPT tubes. These samples will be maintained at room temperature until they are transported to the laboratory.
  Persistence of B-Cell response to Influenza will be measured on study days 0, 7, 28, 90, and 365, and compared for changes.
  Persistence of B-Cell response to Influenza in blood will be measured on study days 0, 7, 28, 90, and 365, and compared for changes.
Changes in Bone marrow persistence of B-Cell response to Influenza | Study Days 0, 28, 365
  Bone marrow aspirate specimens will be drawn, labeled, and logged at the Georgia Clinical & Translational Science Alliance (CTSA) by the Principal Investigator. These samples will be collected in 10 ml sodium heparin tubes and labeled with coded subject information. They will be maintained at room temperature until they are transported to the laboratory.
  Persistence of B-Cell response to Influenza in bone marrow, will be measured on study days 0, 28, and 365, and compared for changes.

CONTACTS AND LOCATIONS:
Overall Officials: Edmund K Waller, MD, PhD, Principal Investigator — Emory University
Locations (1):
- Emory University Hospital, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified genomic data and de-identified health information will be shared
Supporting Information: Study Protocol, ICF
Time Frame: Immediately following publication, no end date
Access Criteria: Researchers who apply for and receive permission to use the information for a specific research project, regarding any research question by controlled-access databases